CLINICAL TRIAL: NCT01946269
Title: Goal-directed Resuscitation in High-risk Patients Undergoing Major Cancer Surgery: a Controlled and Randomized Study
Brief Title: Goal-Directed Therapy in Cancer Surgery
Acronym: GRICS II
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Ludhmila Abrahão Hajjar, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GRICS-02
Record Dates: First submitted 2013-09-16; First posted 2013-09-19 (Estimated); Last update posted 2013-09-19 (Estimated); Status verified 2013-09

CONDITIONS: Postoperative Care
MeSH Terms: interventions — AIEOP acute lymphoblastic leukemia protocol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard group (Active Comparator)
  Interventions: Other: Standard protocol
- Goal-directed therapy (GDT) protocol (Active Comparator)
  Interventions: Other: Goal-directed Resuscitation Therapy (GDT)

INTERVENTIONS:
Other: Goal-directed Resuscitation Therapy (GDT) — * A target value of a cardiac index (CI) greater than 2.5 L/min/m2 and a mean arterial pressure of 70 mmHg will be sought.
  * The first step will be fluid resuscitation with 200ml aliquots of Lactated Ringer's solution plus human albumin 20% 50 mL whenever the CI is lower than 2.5 L/min/m2. The fluid challenge will be stopped if the CVP rises by more than 4 mmHg during the infusion period or CI increases less than 10%.
  * When the CI is lower than or equal to 2.5L/min/m2 despite of fluid challenge, dobutamine will be initiated with increasing doses up to 20mcg/kg/min.
  * The final step will be red blood transfusion to reach a hematocrit higher than 28%.
  * If necessary, norepinephrine infusion will be used to maintain a mean arterial pressure above 70 mmHg.
  Arms: Goal-directed therapy (GDT) protocol
Other: Standard protocol — The control group will be managed by the surgical ICU staff in the postoperative period according to institutional protocol of hemodynamic monitoring.
  Arms: Standard group

SUMMARY:
The purpose of this study is to determine whether a goal-directed resuscitation therapy within the first 8 hours after major abdominal cancer surgery reduces postoperative complications compared to a standard therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to ICU in immediate postoperatory of major abdominal surgery for cancer treatment
* Age over 18 years-old

Exclusion Criteria:

* Weight under 55 kilograms or over 140 kilograms;
* Contra-indication for invasive hemodynamic monitoring;
* Expected ICU permanence less than 24 hours;
* Active bleeding
* Vasoplegic shock with noradrenaline dose higher than 1mcg/kg/min
* Enrolled in other study
* Refuse to consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-03 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint of death or major postoperative complications | 30 days after randomization
  Death or one of the following complications: stroke, renal failure, respiratory complications, cardiovascular complications, deep wound infection and reoperation for any reason.

SECONDARY OUTCOMES:
Duration of ICU stay and hospital stay | 30 days after randomization
  To compare the number of days of ICU stay and hospital stay between groups.
Tissue hypoperfusion markers | 7 days after randomization
  To compare levels of DO2, lactate, ScvO2, base excess and venous to arterial carbon dioxide difference between groups.
Daily SOFA score | 7 days after randomization
  Daily sequential organ failure assessment score within the first 7 days after randomization
Cardiovascular complications | 30 days after randomization
  To compare the incidence of cardiovascular complications between groups. Cardiovascular complications will be defined as myocardial ischemia, acute decompensated heart failure, mesenteric ischemia, pulmonary thromboembolism and peripheral vascular ischemia.
Respiratory complications | 30 days after randomization
  Respiratory complication will be defined as acute distress respiratory syndrome according to Berlin criteria
Severe Renal complication | 30 days after randomization
  Severe renal complication will be defined as renal failure according to Acute Kidney Injury Network (AKIN) stage 3.
Neurological complications | 30 days after randomization
  To compare the incidence of stroke between groups within 30 days after randomization.
Severe infectious complications | 30 days after randomization
  To compare the incidence, between groups, of infectious complications defined as a new septic shock.
Surgical complications | 30 days after randomization
  To compare the incidence between groups of surgical complication. Surgical complication will be defined as reoperation due to any reason, hospital readmission or death

CONTACTS AND LOCATIONS:
Locations (1):
- Intensive Care Unit of the Cancer Institute of Sao Paulo State, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Gerent ARM, Almeida JP, Fominskiy E, Landoni G, de Oliveira GQ, Rizk SI, Fukushima JT, Simoes CM, Ribeiro U Jr, Park CL, Nakamura RE, Franco RA, Candido PI, Tavares CR, Camara L, Dos Santos Rocha Ferreira G, de Almeida EPM, Filho RK, Galas FRBG, Hajjar LA. Effect of postoperative goal-directed therapy in cancer patients undergoing high-risk surgery: a randomized clinical trial and meta-analysis. Crit Care. 2018 May 23;22(1):133. doi: 10.1186/s13054-018-2055-4. PMID 29792232